CLINICAL TRIAL: NCT03440242
Title: Biomarker Discovery in Two Daily Disposable Contact Lenses
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-5982
Record Dates: First submitted 2018-01-25; First posted 2018-02-22 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Visual Acuity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- JJVC Contact Lens (Asymptomatic): Subjects between the ages of 18 and 45 years of age will be enrolled to the JJVC Contact Lens arm based on their habitual lenses and then stratified to an Asymptomatic group based on wear time responses during the baseline assessment.
  Interventions: Device: JJVC Contact Lens
- JJVC Contact Lens (Symptomatic): Subjects between the ages of 18 and 45 years of age will be enrolled to the JJVC Contact Lens arm based on their habitual lenses and then stratified to a Symptomatic group based on wear time responses during the baseline assessment.
  Interventions: Device: JJVC Contact Lens
- Marketed Contact Lens (Asymptomatic): Subjects between the ages of 18 and 45 years of age will be enrolled to the Marketed Contact Lens arm based on their habitual lenses and then stratified to an Asymptomatic group based on wear time responses during the baseline assessment.
  Interventions: Device: Marketed Contact Lens
- Marketed Contact Lens (Symptomatic): Subjects between the ages of 18 and 45 years of age will be enrolled to the Marketed Contact Lens arm based on their habitual lenses and then stratified to a Symptomatic group based on wear time responses during the baseline assessment.
  Interventions: Device: Marketed Contact Lens

INTERVENTIONS:
Device: JJVC Contact Lens — etafilcon A with PVP DD
  Groups: JJVC Contact Lens (Asymptomatic); JJVC Contact Lens (Symptomatic)
Device: Marketed Contact Lens — nelfilcon A DD
  Groups: Marketed Contact Lens (Asymptomatic); Marketed Contact Lens (Symptomatic)

SUMMARY:
This is a non-masked, non-randomized, stratified, 4-arm parallel group, non-interventional study where subjects will be enrolled into one of four arms based on their habitual contact lenses. Subjects will be wearing their habitual contact lenses throughout the study and will be scheduled for morning and afternoon visits totaling 10 visits with a ~4-week washout period between visits 6 and 7.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Appear able and willing to adhere to a no lens wear period of at least one month.
  4. Between 18 and 45 (inclusive) years of age at the time of screening.
  5. Subject must be currently wearing one of the two habitual contact lenses in both eyes (1DAM or DACP) for at least three months. Habitual CL wear is defined as having a minimum wearing time of 3 hours per day, minimum of 3 days per week for at least 3 months.
  6. Subject must have visual acuity of at least 20/40 or better in each eye with their habitual lenses
  7. Subjects must meet one of the following criteria in order to be classified as either asymptomatic or symptomatic group:

     1. Asymptomatic group: CLDEQ-8 score of ≤7, difference between CWT and AWT <1 hours/day
     2. Symptomatic group: CLDEQ-8 score of ≥15, difference between CWT and AWT >3 hours/day
  8. Have healthy eyes with no evidence of abnormality or disease (i.e., no active ocular pathological conditions/ infections of any type).
  9. Have a pair of spectacles that provide corrected binocular visual acuity of 20/40 or better. If no spectacles, subjects must have un-aided binocular visual acuity of 20/40 or better.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating
  2. Any systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
  3. Unacceptable lens fit with their habitual lenses in either eye based on study investigators judgment.
  4. Any extended wear modality.
  5. Use of systemic medications (e.g., chronic steroid use, immuno-suppressants or anti-infective medications) that are known to interfere with contact lens wear.
  6. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
  7. Any previous, or planned (during the course of the study) intraocular/refractive surgery.
  8. Any Grade 3 or 4 slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, and conjunctival injection) on the FDA scale.
  9. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that would contraindicate contact lens wear.
  10. Participation in any interventional contact lens, eye drop or lens care product clinical trial within 30 days prior to study enrollment.
  11. Suspicion of or recent history of alcohol or substance abuse, serious mental illness, or seizures.
  12. Employee of clinical site (e.g., Investigator, Coordinator, Technician).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Summary of Protein (Lysozyme) in Tears | Approximately 2 hours duration of assessment time
  Summarizing potential differences in biomarker responses in tears of subjects wearing two different materials of daily disposable contact lenses. Lysozyme as biomarker in tears will be collected via Schirmer's strips and Capillary tubes at all scheduled visits and will be analyzed using Chromatography.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Narayana Nethralaya Foundation, Bangalore
  - Medical Research Foundation, Chennai